CLINICAL TRIAL: NCT01600430
Title: Early Vitamin D Supplementation for Prevention of Respiratory Morbidity in Extremely Preterm Infants: A Randomized Clinical Trial
Brief Title: Vitamin D Supplementation for Extremely Preterm Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Health System, Alabama (Other)
Responsible Party: Principal Investigator, Namasivayam Ambalavanan, Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UAB Neo 006
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Vitamin D Deficiency; Preterm Infants; Bronchopulmonary Dysplasia
Keywords: Vitamin D; Newborn; Preterm; Supplementation; Respiratory
MeSH Terms: conditions — Vitamin D Deficiency; Bronchopulmonary Dysplasia; Premature Birth | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral Vitamin D--200 IU/day (Active Comparator): Cholecalciferol 200 IU given orally once per day
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (Placebo Comparator): Identical-appearing treatment that does not contain the test drug given orally four times per day.
  Interventions: Dietary Supplement: Placebo
- Oral Vitamin D--800 IU/day (Active Comparator): Cholecalciferol 800 IU given orally once per day
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 200 IU/day given orally once per day as one of 4 doses of 0.5ml each given every 6 hours. Other 3 doses will be placebo (sterile water). Duration of 28 postnatal days
  Other Names: Vitamin D
  Arms: Oral Vitamin D--200 IU/day
Dietary Supplement: Cholecalciferol — 800 IU/day given orally per day as 4 doses of 200 IU/0.5ml each every 6 hours. Duration of 28 postnatal days
  Other Names: Vitamin D
  Arms: Oral Vitamin D--800 IU/day
Dietary Supplement: Placebo — Sterile water 0.5ml given orally every 6 hours. Duration of 28 postnatal days
  Arms: Placebo

SUMMARY:
The study hypothesis states that giving early enteral Vitamin D supplementation to preterm infants will decrease respiratory morbidity in extremely preterm infants.

DETAILED DESCRIPTION:
After informed consent obtained, infants will be randomized using computer-generated stratified randomization codes by the pharmacy. Clinicians, researcher, and primary caregivers will be masked. Subjects will be randomly assigned to one of the treatment arms or to a placebo concurrent control.

Early vitamin D supplementation/placebo will be initiated within the first 7 days after birth. Premature infants will be randomized to receive one of the 3 fixed doses of vitamin D: either placebo (zero dose), 200 IU/day, or 800 IU/day. The supplementation will be started within 72 hours of enteral feeds being initiated and will continue until postnatal day 28. After this period of supplementation, routine supplementation will be conducted in all groups.

Remnant cord blood samples will be analyzed for vitamin D levels (serum hydroxyvitamin D [25(OH)D]. Two circulating vitamin D concentrations (25(OH)D concentrations) will be measured on postnatal days 14 and 28. Urine samples will be collected weekly, to determine calcium excretion if high serum calcium concentrations are found.

Supplementation will be discontinued and infant will exit the study if surgical necrotizing enterocolitis/bowel perforation is diagnosed, if 25 (OH)D concentrations >60ng/mL (>150nmol/L; potentially toxic) are detected or, if infant NPO for greater than 24 hours. If infant made briefly NPO (<24h) for feeding intolerance, suspected sepsis, hypotension,hemodynamically significant PDA, or respiratory difficulties, enteral vitamin D will not be discontinued.

All infants will be followed to discharge for primary, secondary outcomes as well as adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the Regional Newborn ICU of the University of Alabama with gestational age between 23-27 completed weeks

Exclusion Criteria:

* Major congenital/chromosomal anomalies
* Moribund infant with low likelihood of survival, in opinion of the clinical team

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total number of days alive and off respiratory support in the first 28 days | 28 days
  The total number of days alive and off respiratory support. Respiratory support is defined as need of supplemental oxygen and/or positive pressure ventilation to maintain normal target oxygen saturations (88-95%).
Serum vitamin D concentration | Day after birth 28
  Serum vitamin D levels determined by enzyme immunoassay obtained from whole blood (remnant sample or obtained during clinical blood draw)

SECONDARY OUTCOMES:
Number of sepsis episodes treated with antibiotics for at least 5 days | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Number of episodes of culture proven or clinically suspected sepsis episodes treated with antibiotics for at least 5 days
Sepsis | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Culture proven or culture negative clinically treated course consistent with sepsis
Need for supplemental oxygen at 36 weeks of corrected age (Physiologic definition) | 36 weeks gestational age corrected
  A physiologic oxygen challenge test will be administered to infants from 36.0 weeks gestation to 37.0 weeks gestation to determine a need for supplemental oxygen to keep saturation levels between 88-95%.
Duration of mechanical ventilation after randomization | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Counted as number of days on which an infant is on mechanical ventilation for any part of a calendar day
Days alive and off mechanical ventilation in the first 28 days after birth | 28 days
  Counted as days alive without mechanical ventilation for any part of a day
Number of re-intubation events | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Counted as number of reintubations for purposes of respiratory support
Death | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Cardiorespiratory failure
Surgical necrotizing enterocolitis or intestinal perforation | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Radiographic documentation of pneumatosis or intestinal perforation or treatment course for clinical necrotizing enterocolitis per Bell's stage greater than 1.
25(OH)D concentrations >60ng/ml (150 nmol/L) | 14 postnatal (+/- 2 days)
  Vitamin D measurement per blood obtained either centrally or by heel stick.
25(OH)D concentrations >60ng/ml (150 nmol/L) | 28 days postnatal age (+/- 3 days)
  Vitamin D measurement per blood obtained either centrally or by heel stick.
Serum calcium level | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Serum calcium measurement per blood obtained either centrally or by heel stick, performed for clinical care. High serum calcium level is greater than 3 mmol/l of total calcium or total calcium of >12 mg/dL, or ionized calcium >2 mml/L.
Urine calcium level | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Calcium measurement per urine, random sampling. High level (>95%tile) urine calcium to creatinine ratio is >3.8 mmol/mmol.
Meningitis | Participants will be followed for the duration of hospital stay, an expected average of 4 months
  Culture proven or culture negative clinically treated course consistent with meningitis

OTHER OUTCOMES:
Death or Neurodevelopmental Impairment | Birth to 22-26 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Namasivayam Ambalavanan, MD, Principal Investigator — University of Alabama at Birmingham; Ariel A. Salas, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Aristizabal N, Holder MP, Durham L, Ashraf AP, Taylor S, Salas AA. Safety and Efficacy of Early Vitamin D Supplementation in Critically Ill Extremely Preterm Infants: An Ancillary Study of a Randomized Trial. J Acad Nutr Diet. 2023 Jan;123(1):87-94. doi: 10.1016/j.jand.2022.06.012. Epub 2022 Jun 18. PMID 35728797
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Fort P, Salas AA, Nicola T, Craig CM, Carlo WA, Ambalavanan N. A Comparison of 3 Vitamin D Dosing Regimens in Extremely Preterm Infants: A Randomized Controlled Trial. J Pediatr. 2016 Jul;174:132-138.e1. doi: 10.1016/j.jpeds.2016.03.028. Epub 2016 Apr 11. PMID 27079965